CLINICAL TRIAL: NCT03845972
Title: Effect of Ultrasound-guided Saphenous Nerve and Nerve to Vastus Medialis Block Within Subsartorial Femoral Triangle on Quadriceps Strength
Brief Title: Effect of Saphenous Nerve and Nerve to Vastus Medialis Block Within Subsartorial Femoral Triangle on Quadriceps Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Alisa Seangleulur, Assistant Professor, Thammasat University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ทป.2/44/2561
Record Dates: First submitted 2019-01-19; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Saphenous Nerve Block; Regional Anesthesia Morbidity; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- before SSFTB (No Intervention)
- after SSFTB (Experimental)
  Interventions: Procedure: SSFTB

INTERVENTIONS:
Procedure: SSFTB — Patients who underwent major knee surgery and had already planned to perform subsartorial femoral triangle block (SSFTB) were included in the study. They were measured the outcomes the night before surgery. The saphenous nerve and nerve to vastus medialis were blocked at the subsartorial femoral triangle level by experienced anesthesiologists. After standard monitor, the distal femoral triangle was identified 2 cm proximal to the opening of adductor canal by ultrasound guidance. At this level, The location of nerve to vastus medialis was confirmed by nerve stimulator and it was blocked with 0.5% levobupivacaine 5 ml. Then, 0.5% levobupivacaine 10 ml would be injected perifemoral artery. The outcomes were re-assessed 30 min after block.
  Other Names: nerve to vastus medialis and saphenous nerve block
  Arms: after SSFTB

SUMMARY:
This research objective is to compare quadriceps strength by measuring maximal voluntary isometric contraction (MVIC) and risk of fall before and after subsartorial femoral triangle block (SSFTB)

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are all ASA class I-III, age 18-80 years, and have plan to perform SSFTB at Thammasat University Hospital consecutively

Exclusion Criteria:

* Exclusion criteria are patients who refuse to participate the study, morbid obesity (BMI ≥ 35 kg.m2), lower extremity neurological dysfunction, performing other peripheral nerve blocks, patients who cannot cooperate or measure MVIC, difference of quadriceps strength between two side of knees more than 10 percent, and SSFTB is not finally performed or failed block.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
quadriceps strength | 30 minutes after SSFTB
  Quadriceps strength will be assessed as MVIC with handheld dynamometer (HHD, Lafayette Instrument, Lafayette, IN).

SECONDARY OUTCOMES:
motor power of knee extension | 30 minutes after SSFTB
  The muscle power will be graded compared to another leg: 0 = No motor block, 1 = partial motor block, 2 = complete motor block.
perception of fall 30 minutes | 30 minutes after SSFTB
  If the patient can be able to stand independently for at least 30 seconds without support, he or she will be asked to do functional reach test, which the patient should reach forward by staying put feet. The difference of starting and ending point of the reaching hand will be measured. If the patient cannot stand independently for at least 30 seconds without support or do functional reach test less than 25 cm indicates that he or she has a higher risk for falls.

CONTACTS AND LOCATIONS:
Locations (1):
- Ratibhorn Rangsee, Klong Luang, Pratumthani, Thailand

IPD SHARING:
Plan to Share IPD: No